CLINICAL TRIAL: NCT04559464
Title: Fissure Closure With the AeriSeal System for CONVERTing Collateral Ventilation Status in Patients With Severe Emphysema; A Multicenter, Prospective Trial
Brief Title: Fissure Closure With the AeriSeal System for CONVERTing Collateral Ventilation Status (CONVERT)
Acronym: CONVERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pulmonx Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 630-0030-01
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Emphysema; COPD; Severe Emphysema
Keywords: Bronchoscopic lung volume reduction; Zephyr Valves; AeriSeal
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive | interventions — Pneumonectomy

STUDY DESIGN:
Intervention Model Description: Stage 1 will address the closure of the lobar fissure gaps (or collateral air channels) to block collateral ventilation (CV) with the AeriSeal System (conversion of the CV+ target lobe to CV-). Stage 2 will include successfully converted subjects in Stage 1. Converted CV- target lobes will follow standard of care and receive the Zephyr Endobronchial valves per the Zephyr Instructions for Use (IFU) to perform bronchoscopic lung volume reduction (BLVR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AeriSeal and Zephyr Valve Treatment (Other): Stage 1 will address the closure of the lobar fissure gaps (or collateral air channels) to block collateral ventilation (CV) with the AeriSeal System (conversion of the CV+ target lobe to CV-).
  Stage 2 will include successfully converted subjects in Stage 1. Converted CV- target lobes will follow standard of care and receive the Zephyr Endobronchial valves per the Zephyr Instructions for Use (IFU) to perform bronchoscopic lung volume reduction (BLVR).
  Interventions: Device: AeriSeal; Device: Zephyr Valves

INTERVENTIONS:
Device: AeriSeal — The AeriSeal Foam functions by blocking both small airways and collateral channels causing absorption atelectasis in the treated region of the lung. Occlusion with the foam also yields a targeted fibrotic response which durably reduces lung hyperinflation. The reduction in hyperinflation allows the healthier parts of the lung to re-inflate and improve breathing mechanics and gas exchange. In this study, the AeriSeal delivery will be limited to three segments that contain the collateral channel(s) between lung lobes. A minimum 10 mL volume of AeriSeal will be delivered per segment, with a total delivered volume limit of 40 mL per subject (including re-treatment, if needed) in a total of three segments.
Device: Zephyr Valves — The Zephyr Valves are implantable bronchial valves intended to control airflow in order to improve lung function in patients with hyperinflation associated with severe emphysema and/or to reduce air leaks.
  Other Names: Bronchoscopic Lung Volume Reduction (BLVR); Zephyr System

SUMMARY:
This is a prospective, open-label, multi-center, single-arm study to be conducted at up to 20 investigational sites. The Study plans to enroll up to 140 subjects with severe emphysema and collateral ventilation in the target lobe. This protocol is designed to evaluate the utility of the AeriSeal System to occlude collateral air channels in a target lung lobe with collateral ventilation (CV) and convert the target lung lobe to having little to no collateral ventilation. Subjects can then receive Zephyr Valves to achieve atelectasis in the targeted lobe, once AeriSeal has converted the CV+ lobe to a CV- one. Therefore, the study will have two Stages:

• Stage 1 will address the closure of the lobar fissure gaps (or collateral air channels) to block collateral ventilation (CV) with the AeriSeal System; conversion of the CV+ target lobe to CV-. Conversion of collateral ventilation will be evaluated by Chartis after 45 days. In the case of unsuccessful conversion, a second treatment of AeriSeal may be attempted, provided that the total application volume from both the initial and the repeat treatments does not exceed 40 mL in up to three (3) segments.

Clinical Assessments post-AeriSeal will be conducted at 28 and 45 days after first treatment and repeated after the second treatment, if applicable. For the purpose of protocol follow-up, the Day 45 post-AeriSeal final treatment will equal Day 0 for Stage 2.

• Stage 2 will include successfully converted subjects; CV+ to CV- conversion in Stage 1. Converted CV- target lobes will follow standard of care and receive CE marked Zephyr Endobronchial valves per the Zephyr IFU to perform bronchoscopic lung volume reduction (BLVR).

Clinical assessments will be conducted at 45 Days, 3-months, 6-months, and 12-months post-Zephyr Valve procedure.

DETAILED DESCRIPTION:
Severe emphysema subjects will be consented using an Ethics Committee approved Informed Consent Form (ICF) for baseline evaluations. Subjects with ≥ 50% lobar emphysema destruction (evaluated quantitatively by using percentage lung volume occupied by low-attenuation regions/voxels) and identified as potentially having collateral ventilation, with fissure completeness ≥ 80% from the Quantitative Computed Tomography (QCT) report (CV status later to be confirmed by Chartis assessment at Visit 2) will undergo additional QCT assessment for the feasibility of directing AeriSeal to the appropriate segment to seal the anatomical defect. Subjects in whom this is considered feasible will be enrolled.

Enrolled subjects will undergo a bronchoscopy procedure during which the presence of collateral ventilation will be confirmed using the Chartis Pulmonary Assessment System (Pulmonx Corporation) and if confirmed, will undergo AeriSeal treatment in the segment(s) feeding the collateral channel. A minimum 10 mL volume of AeriSeal will be delivered per segment, with a total delivered volume limit of 40 mL per subject (including re-treatment, if needed) in a total of three segments. Subjects will be hospitalized for a minimum of two (2) nights for observation and discharged if stable. Following discharge, subjects will be contacted daily for at least 7 days via telephone to assess status and solicit any Adverse Events.

Subjects that have little to no collateral ventilation at the initial bronchoscopy, as assessed by the Chartis Pulmonary Assessment System, will be exited from the study.

Six (6) weeks following the AeriSeal treatment, subjects will undergo a second bronchoscopy procedure for assessment of collateral ventilation status of the AeriSeal treated lobe with Chartis. If the Chartis assessment shows presence of collateral ventilation (CV+) at the lobar level, Chartis will be used to assess collateral ventilation at the segmental level to identify the segment with open collaterals. A second treatment with AeriSeal will be considered, provided the total delivered volume inclusive of the original treatment does not exceed 40 mL per subject. The post-procedure follow-up assessments for the second treatment will be repeated as after the initial treatment.

If the Chartis assessment determines little to no collateral ventilation (CV-) in the AeriSeal treated lobe, the lobe will be treated with Zephyr Valves as per the standard valve placement procedure. Subject will be hospitalized for a minimum of three (3) nights post-valve placement procedure and discharged with follow-up in accordance with this protocol, which includes standard post-valve placement follow-up.

Subjects who do not convert from CV+ to CV- status will continue to be observed for safety through 12 months following AeriSeal treatment or re-treatment, whichever is later.

The primary AeriSeal endpoint is the percentage of study subjects that are successfully converted from a positive collateral ventilation (CV+) status in the treated lobe to having little to no collateral ventilation (CV-) in the treated lobe.

Following the procedure for Zephyr Valve placement, subjects will be required to undergo Pulmonary Rehabilitation as per the local/national guidelines of each participating institution; at least 20 supervised sessions. A High Resolution Computed Tomography (HRCT) will be performed at 45-days post-Zephyr Valve procedure to determine Treated Lobe Volume Reduction (TLVR). Lung function will be assessed by measuring post-bronchodilator FEV1. A valve adjustment procedure will be considered if there is lack of TLVR (≤ 350 mL reduction from the pre-valve assessment) following evaluation of the High-resolution computed tomography (HRCT) to determine which valve needs to be replaced or addition of a new valve at a previously missed airway. Subjects will also be evaluated at 3-months, 6-months, and 12 months following Zephyr Valve placement.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is willing and able to provide Informed Consent and to participate in the study.
2. Subject is ≥ 40 and ≤ 75 years of age at the time Informed Consent signature.
3. Subject has at least one lobe with ≥ 50% emphysema destruction (at -910 HU) as determined by QCT.
4. Subject has a diagnosis of homogenous or heterogeneous emphysema, confirmed by HRCT scan. Heterogeneous emphysema defined as ≥ 15% difference (at -910 HU) in emphysema destruction score of adjacent lobes by HRCT.
5. Subject has a gap in the interlobar fissure that corresponds to one or more segments as determined by QCT.
6. Subject has clinically significant dyspnea with a mMRC Dyspnea score ≥ 2.
7. Subject has a Six-Minute Walk Distance ≥ 250 meters.
8. Subject has post-bronchodilator FEV1 ≥ 15% predicted and ≤ 50% predicted.
9. Subject has post-bronchodilator Total Lung Capacity ≥ 100% predicted.
10. Subject has post-bronchodilator Residual Volume ≥ 150% predicted if heterogeneous emphysema and ≥ 200% predicted if homogeneous emphysema.
11. Subject has stopped smoking for at least eight (8) weeks prior to Screening visit as confirmed by carboxyhemoglobin or cotinine levels.
12. Subject has received preventive vaccinations against potential respiratory infections consistent with local recommendations or policy.

Exclusion Criteria:

1. Subject has severe bullous emphysema where bulla is ≥ 1/3 of the total lung volume.
2. Subject has had prior lung volume reduction surgery, prior lobectomy or pneumonectomy, prior lung transplantation, prior airway stent placement, prior ipsilateral pleurodesis, or prior endobronchial lung volume reduction therapy of any type.
3. Subject has evidence of active respiratory infection.
4. Subject has an ongoing COPD exacerbation or bronchospasm.
5. Subject has a known allergy to the device components:

   1. Polyether block amide - PEBAX®
   2. Polyvinyl Alcohol
   3. Glutaraldehyde
   4. Nitinol (nickel-titanium) or its constituent metals (nickel or titanium)
   5. Silicone
6. Subject requires invasive ventilatory support (NOTE: The use of continuous Positive Airway Pressure (CPAP) and BiPAP devices for Sleep Apnea is permitted).
7. Subject has post-bronchodilator Diffusion Capacity (DLCO) < 20% predicted.
8. Subject cannot tolerate corticosteroids or relevant antibiotics.
9. Subject has other relevant comorbidities as judged by the Investigator or is deconditioned and cannot tolerate the stress of post-treatment inflammatory response.
10. Subject has had three (3) or more COPD exacerbations requiring hospitalization during the year prior to Informed Consent signature.
11. Subject has severe gas exchange abnormalities as defined by any one of the following (test conducted at rest on room air as tolerated, or on up to 4 L/min supplemental O2):

    1. PaCO2 ≥ 55 mm Hg (7.3 kPa)
    2. PaO2 < 45 mm Hg (6.0 kPa)
    3. SpO2 < 90%
12. Subject has uncontrolled pulmonary hypertension, defined as peak pulmonary systolic pressure > 45 mm Hg on echocardiogram or right heart catheterization.
13. Subject use of systemic steroids > 20 mg/day prednisolone or equivalent within 4 weeks of Informed Consent signature.
14. Subject use of immunosuppressive agents within four (4) weeks of Informed Consent signature.
15. Subject whose use heparins and oral anticoagulants (e.g., warfarin, dicumarol) cannot be discontinued according to local pre-procedural protocols. Note: antiplatelet drugs including aspirin and clopidogrel are permitted.
16. Subject's CT scan indicates the presence of any the following radiologic abnormalities:

    1. Pulmonary nodule on CT scan greater than 0.8 cm in diameter (Does not apply if present for one (1) year or more without increase in size or if proven benign by biopsy).
    2. Radiologic picture consistent with active pulmonary infection, e.g., unexplained parenchymal infiltrate.
    3. Significant interstitial lung disease.
    4. Significant pleural disease.
17. Subject's baseline EKG indicates non-atrial arrhythmias or conduction abnormalities.
18. Subject has high cardiac risk after undergoing cardiac risk assessment in accordance with published guidelines or ischemic heart disease, congestive heart failure, renal failure, or cerebrovascular disease.
19. Subject has clinically significant asthma (reversible airway obstruction), chronic bronchitis, or bronchiectasis.
20. Subject has allergy or sensitivity to medications required to safely perform bronchoscopy under conscious sedation or general anesthesia.
21. Subject participated in an investigational study of a drug, biologic, or device not currently approved for marketing within 30 days prior to Screening visit. Subjects being followed as part of a long-term surveillance of a non-pulmonary study that has reached its primary endpoint are eligible for participation in this study.
22. Subject has Body Mass Index (BMI) < 18 kg/m2 or > 35 kg/m2.
23. Subject is a female who is pregnant, breast-feeding, or planning to be pregnant in next 12 months.
24. Subject has clinically significant abnormal screening laboratory test results per the Institution specific reference laboratory normal values for the following:

    1. White blood cells (total)
    2. Hematocrit
    3. Platelets
    4. Prothrombin time or INR
    5. Partial thromboplastin time
    6. Positive β-HCG Pregnancy test (if female)
25. Subject has evidence of severe disease which in the judgment of the Investigator may compromise survival for the duration of the study (at least 12 months) e.g.:

    1. HIV/AIDs
    2. Active malignancy
    3. Stroke or Transient Ischemic attack (TIA) within 12 months of Screening visit
    4. Myocardial infarction within six (6) months of the Screening visit
    5. Congestive heart failure within six (6) months of the Screening visit defined as clinical evidence of right or left heart failure or left ventricular ejection fraction < 45% on echocardiogram
26. Subject has uncontrolled diabetes mellitus.
27. Subject has any other condition that the Investigator believes would interfere with the intent of the study or would make participation not in the best interest of the subject including but not limited to alcoholism, high risk for drug abuse, or noncompliance in returning for follow-up visits.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects converted from a positive collateral ventilation status (CV+) to having little to no collateral ventilation (CV-) in the treated lobe. | 6-weeks post-AeriSeal treatment
  The primary AeriSeal endpoint will be the percentage of study subjects that are successfully converted from a positive collateral ventilation status (CV+) in the treated lobe to having little to no collateral ventilation (CV-) in the treated lobe six (6) weeks after delivery of AeriSeal.
Treated Lobe Volume Reduction (TLVR) responders | 45-days post-Zephyr Valve treatment
  The primary Zephyr Valve endpoint is the percentage of subjects achieving TLVR ≥ 350 mL (TLVR Responders) at 45-days post-valve treatment. That is, the percentage of CV+ to CV- converted subjects from Stage 1 who subsequently receive valves and have Treated Lobe Volume Reduction (TLVR) of ≥ 350 mL, via High-resolution computed tomography (HRCT) at 45-days post-valve treatment.

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 3-months
  Post-Bronchodilator Forced Expiratory Volume in 1 second (FEV1) change from Baseline to 3-months (Absolute and Percent changes)
Residual volume (RV) | 3-months
  Residual volume (RV) change from Baseline to 3-months (Absolute and Percent changes).

OTHER OUTCOMES:
Forced Expiratory Volume in 1 second (FEV1) | 6-months and 12-months
  Post-Bronchodilator Forced Expiratory Volume in 1 second (FEV1) change from Baseline to 6-months and 12-months (Absolute and Percent changes)
Residual volume (RV) | 6-months and 12-months
  Residual volume (RV) change from Baseline to 6-months and 12-months (Absolute and Percent changes).
Six-Minute Walk Distance (6MWD) | 3-months, 6-months, and 12-months
  Change in Six-Minute Walk Distance (6MWD) from Baseline to 3-months, 6-months, and 12-months.
St. George's Respiratory Questionnaire (SGRQ) Total Score | 3-months, 6-months, and 12-months
  Change in St. George's Respiratory Questionnaire (SGRQ) Total Score from Baseline to 3-months, 6-months, and 12-months.
  The St. George's Respiratory Questionnaire measures health status (quality of life) in patients with diseases of airways obstruction. Scores range from 0 to 100, with higher scores indicating more limitations.
Modified Medical Research Council Dyspnea Score (mMRC) | 3-months, 6-months, and 12-months
  Change in the Modified Medical Research Council (mMRC) Dyspnea Scale from Baseline to 3-months, 6-months, and 12-months.
  The mMRC (Modified Medical Research Council) stratifies severity of dyspnea in respiratory diseases. The severity of dyspnea is rated on a scale of 0 to 4, with higher scores indicating more limitations.
Total Lung Capacity (TLC) | 3-months, 6-months, and 12-months
  Changes in TLC from Baseline to 3-months, 6-months, and 12-months (Absolute and Percent changes).
Inspiratory Capacity (IC) | 3-months, 6-months, and 12-months
  Changes in IC from Baseline to 3-months, 6-months, and 12-months (Absolute and Percent changes).
Residual Volume/Total Lung Capacity (RV/TLC) ratio | 3-months, 6-months, and 12-months
  Changes in the RV/TLC ratio from Baseline to 3-months, 6-months, and 12-months (Absolute and Percent changes).
Inspiratory Capacity/Total Lung Capacity (IC/TLC) ratio | 3-months, 6-months, and 12-months
  Changes in the IC/TLC ratio from Baseline to 3-months, 6-months, and 12-months (Absolute and Percent changes).
Treated Lobe Volume Reduction (TLVR) | 6-months and 12-months
  Changes in TLVR from Baseline to 6-months and 12-months.

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Percy, Study Director — Pulmonx Corporation
Locations (14):
- Australia (2):
  - The Wesley Hospital, Brisbane
  - Macquarie University Hospital, Sydney
- France (2):
  - CHU Limoges, Limoges
  - CHU Toulouse, Toulouse
- Germany (3):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Ruhrlandklinik Essen, Essen
  - ThoraxKlinik, Heidelberg
- ASST Spedali Civili, University Hospital, Brescia, Italy
- University Medical Center Groningen, Groningen, Netherlands
- University Hospital of Zurich, Zurich, Rämistrasse 100, Switzerland
- United Kingdom (4):
  - Golden Jublilee National Hospital, Clydebank, Scotland
  - University Hospital of Wales, Cardiff
  - Royal Brompton Hospital, London
  - Nottingham University Hospitals, Nottingham

IPD SHARING:
Plan to Share IPD: No